CLINICAL TRIAL: NCT02008448
Title: Endomyocardial Botulinum Toxin Injection in Patients With Persistent Atrial Fibrillation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT_AFPers
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI+LL (Active Comparator): Circumferential PVI was accomplished and then additional ablation lines were created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the LA between the two superior PVs (roof). Finally, patients underwent cavo-tricuspid isthmus ablation in the right atrium.
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Linear Lesion Ablation
- PVI+LL+BT injection (Active Comparator): Circumferential PVI was accomplished and then additional ablation lines were created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the LA between the two superior PVs (roof). Finally, patients underwent cavo-tricuspid isthmus ablation in the right atrium.
  Injection of the botulinum toxin is performed in main anatomical zones of ganglionated plexuses of left atrium using Myostar catheter (Biosense Webster).
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Linear Lesion Ablation; Drug: BT injection

INTERVENTIONS:
Procedure: Pulmonary vein isolation
Procedure: Linear Lesion Ablation
Drug: BT injection
  Arms: PVI+LL+BT injection

SUMMARY:
The investigators have conducted a prospective, double-blind, randomized study to assess the comparative safety and efficacy of two different ablation strategies, PVI plus linear lesions (LL) plus botulinum toxin injection versus PVI plus linear lesions (LL), in patients with persistent or longstanding persistent AF. Results were assessed with the use of an implanted monitoring device (IMD).

ELIGIBILITY:
Inclusion Criteria:

* Persistent and longstanding persistent AF

Exclusion Criteria:

* congestive heart failure
* LV ejection fraction < 35%
* left atrial diameter > 60 mm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
freedom of atrial tachyarrhythmia, including AF and atrial flutter/tachycardia | 1 year

SECONDARY OUTCOMES:
serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- University of Rochester, Rochester, New York, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru